CLINICAL TRIAL: NCT07163234
Title: First-In-Human Study (Phase I) Evaluating the Safety of the IPERF Femoral Arterial Cannula in Patients Undergoing a Planned Cardiac Surgery Requiring the Use of an Extracorporeal Circulation Via a Femoral Approach for a Maximum of 6 Hours
Brief Title: Safety of the IPERF Femoral Arterial Cannula in Patients Undergoing Planned Cardiac Surgery With Extracorporeal Circulation Via Femoral Approach
Acronym: FIH IPERF-01
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IPERF SAS (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IPERF-01
Record Dates: First submitted 2025-08-27; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Surgery; Ischemia Limb
Keywords: Ischemia; Cardiac Surgery
MeSH Terms: conditions — Ischemia | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental): Single arm
  Interventions: Device: Cardiac surgery

INTERVENTIONS:
Device: Cardiac surgery — cardiac surgery

SUMMARY:
This is a first-in-human, prospective, single-arm, phase I clinical study evaluating the safety of the iPerf femoral arterial cannula in patients undergoing planned cardiac surgery requiring extracorporeal circulation (ECC) via a femoral approach for up to 6 hours. The iPerf device is a dual-lumen arterial cannula designed to provide systemic and lower limb perfusion during ECC, with the goal of reducing the risk of acute limb ischemia. The study will be conducted at a single center in France and will include 15 adult patients. Primary outcomes focus on procedure-related and late adverse events up to 30 days post-surgery. Secondary objectives include assessment of ischemic events, tissue oxygen saturation, and surgeon satisfaction with device handling. The study aims to demonstrate feasibility and safety of the iPerf cannula as an innovative solution for lower limb perfusion during femoral artery cannulation.

DETAILED DESCRIPTION:
This is a first-in-human, prospective, single-arm, phase I clinical study evaluating the safety of the iPerf femoral arterial cannula in patients undergoing planned cardiac surgery requiring extracorporeal circulation (ECC) via a femoral approach for up to 6 hours. The iPerf device is a dual-lumen arterial cannula designed to provide systemic and lower limb perfusion during ECC, with the goal of reducing the risk of acute limb ischemia. The study will be conducted at a single center in France and will include 15 adult patients. Primary outcomes focus on procedure-related and late adverse events up to 30 days post-surgery. Secondary objectives include assessment of ischemic events, tissue oxygen saturation, and surgeon satisfaction with device handling. The study aims to demonstrate feasibility and safety of the iPerf cannula as an innovative solution for lower limb perfusion during femoral artery cannulation.

ELIGIBILITY:
Inclusion criteria

* Patient aged 18 years or older
* Patient able to understand the study procedures, provide written informed consent, and comply with study procedures
* Patients with planned cardiac surgery requiring the use of an extracorporeal circulation via a femoral approach for a maximum of 6 hours.
* Patient affiliated to the social security system

Exclusion criteria

* Patient weighting less than 45 kg
* Patient weighting more than 130 kg
* Patient with common femoral artery diameter less or equal to 6 mm
* Patient with a stenosis of the aorta, iliac artery, or femoral artery reducing their diameter of more than 50%
* Patient with previous vascular or endovascular surgery of the iliac or femoral arteries
* Patient participating in another interventional study
* Patients with known arterial dissection
* Patient who is pregnant at the time of enrollment
* Patients under judicial protection, guardianship or curatorship or subjects deprived of their liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety of the novel IPERF femoral arterial cannula | From enrollment to 30-60 days post surgery
  Per procedure and late adverse events related to the IPERF Femoral Arterial Cannula, up to 30 days after surgery.

SECONDARY OUTCOMES:
Number of patients with at least one ischemic event from cannula installation to decannulation | From enrollment to 30-60 days post surgery
  Number of patients with at least one clinical ischemic event from cannula installation to decannulation defined by clinical observations of the cannulated limb: paleness/ bluish appearance of the leg, oedema, coldness and increased skin recolouring time.
Evolution of Tissue Oxygen Saturation (StO2) versus baseline during femoral cannulation with IPerf™ device between the cannulated and the non-cannulated lower limb. | From enrollment to 30-60 days post surgery
  Evolution of Tissue Oxygen Saturation (StO2) versus baseline the cannulated and non cannulated limb (Ceulemans Heart and Vessels, 2023 and versus baseline during femoral cannulation with IPerf™ device in the cannulated and non-cannulated lower limb by NIRS method
Satisfaction of the surgeon | From enrollment to 30-60 days post surgery
  Satisfaction of the surgeon regarding insertion, positioning, stability, and withdrawal of the device: satisfaction score ≥3 (satisfaction scale: 1- Very dissatisfied, 2- Dissatisfied, 3-Neither dissatisfied or satisfied, 4- Satisfied, 5- Very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Mordant, Surgeon, Study Director
Locations (1):
- Hôpital privé Jacques Cartier - Ramsay Santé, Massy, France

IPD SHARING:
Plan to Share IPD: No